CLINICAL TRIAL: NCT02495051
Title: Prevalence of Barrett's Esophagus in Adolescents and Young Adults With Esophageal Atresia
Brief Title: Esophageal Atresia: Metaplasia, Barrett
Acronym: Oesophagix
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/cic; DR-2011-057 / A 910270 (Other: CNIL Number)
Record Dates: First submitted 2015-06-22; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Gastroesophageal Reflux; Esophagus, Barrett
Keywords: gastroesophageal reflux; barrett esophagus
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single group-study
  Interventions: Procedure: esophageal biopsies

INTERVENTIONS:
Procedure: esophageal biopsies

SUMMARY:
The frequency of Barrett's esophagus (BE) has increased in adults in the last decades, but BE is rare in children. Esophageal atresia (EA), the most common congenital anomaly affecting the esophagus, predisposes the patient to severe and prolonged gastroesophageal reflux disease. Because gastroesophageal reflux disease plays a major role in the development of BE by causing repeated mucosal damage, development of BE is a concern even in children and young adults in this specific population. The aim of this study is to assess the prevalence of BE (gastric and/or intestinal metaplasia) in a population of adolescents/young adults who had been treated for EA in early infancy. All eligible patients received upper gastrointestinal endoscopy under general anesthesia with standardized esophageal staged biopsies. Histological suspicion of metaplasia was confirmed centrally.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of esophageal atresia (all types, Ladd's classification)

Exclusion Criteria:

* No medical history of esophageal atresia
* Non acceptance to participate from the patient and/or his parents
* esophageal atresia treated with esophageal replacement (e.g., coloplasty, gastric transposition)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All esophageal atresia patients treated in 20 centers that participated in the French-speaking Group of Gastroenterology, Hepatology, and Nutrition and/or were members of the esophageal atresia national registry
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
presence of gastric and / or intestinal metaplasia diagnosed at histology | during 2 hours of the endoscopy exam
  Prevalence of Barrett's esophagus (gastric and/or intestinal metaplasia) in adolescents treated for esophageal atresia

SECONDARY OUTCOMES:
presence of esophagitis or anomalies at the anastomotic stage diagnosed at histology | during 2 hours of the endoscopy exam
evaluation of the nutritional status | during the single visit scheduled, the day of endoscopy. This periode is corresponding at a day hospitalization (less than 12 hours in the day)
evaluation of actual symptoms and treatment of gastroesophageal reflux disease | during the single visit scheduled, the day of endoscopy. This periode is corresponding at a day hospitalization (less than 12 hours in the day)
evaluation of actual other symptoms (respiratory, dysphagia) | during the single visit scheduled, the day of endoscopy. This periode is corresponding at a day hospitalization (less than 12 hours in the day)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gottrand, MD, PhD, Study Chair — University Hospital, Lille
Locations (20):
- Belgium (4):
  - Cliniques Universitaires St Luc,, Brussels
  - Department of Pediatric Gastroenterology, AZ VUB,, Brussels
  - Department of Pediatric Gastroenterology, HUDERF,, Brussels
  - Department of Gastroenterology CHC, Liège, Liège
- Hôpital Mère-Enfants Ste Justine, Montréal, Canada, Montreal, Canada
- France (14):
  - CHU Angers, Angers
  - CHU, Bordeaux, Bordeaux
  - CHU, Caen, Caen
  - Centre Hospitalier, Le Havre
  - University Hospital, Hôpital Jeanne de Flandres, Lille
  - CHU, Lyon, Lyon
  - CHU, Nantes, Nantes
  - AP-HP ,Hôpital Robert Debré,, Paris
  - AP-HP Hôpital Trousseau, Paris
  - CHU, Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CH Départemental Félix Guyon,, Saint Denis-La Réunion
  - CHU, Strasbourg, Strasbourg
  - CHU Toulouse,, Toulouse
- Centre Hospitalier de Luxembourg,, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Schneider A, Gottrand F, Bellaiche M, Becmeur F, Lachaux A, Bridoux-Henno L, Michel JL, Faure C, Philippe P, Vandenplas Y, Dupont C, Breton A, Gaudin J, Lamireau T, Muyshont L, Podevin G, Viola S, Bertrand V, Caldari D, Colinet S, Wanty C, Sauleau E, Leteurtre E, Michaud L. Prevalence of Barrett Esophagus in Adolescents and Young Adults With Esophageal Atresia. Ann Surg. 2016 Dec;264(6):1004-1008. doi: 10.1097/SLA.0000000000001540. PMID 26720426